CLINICAL TRIAL: NCT03028935
Title: Fuerte y Sanas: Exercise and Nutrition Program in Improving Physical Activity and Dietary Behavior in Non-Active, Overweight, or Obese Latinas
Brief Title: Exercise and Nutrition Program in Improving Physical Activity and Dietary Behavior in Non-Active, Overweight, or Obese Latinas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Cynthia Perry, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00011637; NCI-2016-01321 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB00011637 (Other: OHSU Knight Cancer Institute); P30CA069533 (NIH); R03CA197657 (NIH)
Record Dates: First submitted 2016-09-22; First posted 2017-01-23 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

ARMS (1):
- Prevention (exercise, nutrition education program) (Experimental): Exercise Intervention & Nutritional Intervention. Participants undergo instructor-led exercise and nutrition education classes for 60 minutes twice a week for 12 weeks.
  Interventions: Behavioral: Exercise Intervention; Behavioral: Nutritional Intervention

INTERVENTIONS:
Behavioral: Exercise Intervention — Undergo instructor-led exercise program
Behavioral: Nutritional Intervention — Undergo instructor-led nutritional education program

SUMMARY:
This pilot clinical trial studies how well an evidence-based exercise and nutrition program adapted for Latinas works in improving physical activity and dietary behavior in non-active, overweight, or obese rural Latinas. An exercise and nutrition program may reduce the risk for developing certain cancers, obesity, and chronic health conditions in Latinas who are non-active, overweight, or obese.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Adapt an effective evidence-based exercise and nutrition program to meet the needs of rural Latinas.

II. Implement the adapted program in a rural Latina population. III. Evaluate feasibility and potential to improve physical activity and dietary behavior of the adapted program in a rural Latina population.

OUTLINE:

Phase I: Create a community advisory board to adapt Strong Women Healthy Hearts Program (SWHHP) using feedback on the existing SWHHP from Latinas residing in the community.

Phase II: Conduct a small pilot study to assess effectiveness of the adapted program (one group pre-post design, with data collected at three time points).

INTERVENTION GROUP: Participants undergo instructor-led exercise and nutrition education classes for 60 minutes each twice a week for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Phase I:
* Bilingual Latina
* Live in the community
* Phase II:
* Latina
* Currently non-active (exercise two days or less per week)
* Overweight or obese (body mass index [BMI] of 24 or greater)

Exclusion Criteria:

* A medical condition that precludes moderate-vigorous physical activity as determined by health care provider
* Pregnancy

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-07-05 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2018-03-19 (Actual)

PRIMARY OUTCOMES:
Change in weight | Baseline up to post intervention, up to 7 months
  Mean and standard deviation will be calculated.

SECONDARY OUTCOMES:
Change in fitness level as assessed by the 6 minute walk test | Baseline up to post intervention, up to 7 months
  The distance walked in 6 minutes will be recorded. Mean and standard deviation will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Perry, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States